CLINICAL TRIAL: NCT01571180
Title: Influence of Obesity and Gastric Bypass on Medication Absorption: Prospective Follow-up of Patients
Brief Title: Influence of Obesity and Gastric Bypass on Medication Absorption
Acronym: INOGMA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Ina Gesquiere, Principal Investigator, KU Leuven
Other Study IDs: s53782
Record Dates: First submitted 2012-04-02; First posted 2012-04-05 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Obesity
Keywords: Obesity; Gastric bypass; Medication; Medication counseling; Dietary pattern; Follow-up of patients
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gastric Bypass: Obese patients who have scheduled a gastric bypass

SUMMARY:
Patients who have scheduled a gastric bypass (RYGB) in UZ Leuven, will be questioned preoperatively and one, three, six and twelve months after gastric bypass surgery. The purpose of this study is to explore current practice regarding the use of medication and medication counseling after RYGB and to examine the changes in dietary pattern before and after RYGB.

DETAILED DESCRIPTION:
Target group: patients who have scheduled a gastric bypass in UZ Leuven. Patients will be questioned preoperatively and one, three, six and twelve months after gastric bypass surgery. Each assessment will be performed during a routine consultation.

The following aspects will be investigated:

* Medication The investigators have composed a questionnaire to examine which drugs the patients use, adherence, information received about medication and from whom,…
* Clinical parameters Every consultation, concentrations of hemoglobin, iron, hepcidin, vitamin B12,…. and a 24h urine collection to determine calcium excretion will be collected.
* Dietary intake The investigators will ask patients to keep a food record during two non-consecutive days preceding each consultation. In this food record patients have to note all consumed foods and beverages with the right/estimated amounts. This makes it possible to see the changes of the composition of the meals before and after RYGB.
* Body composition

ELIGIBILITY:
Inclusion Criteria:

* Patients who have scheduled gastric bypass
* Use of at least one chronic drug (including contraception)

Exclusion Criteria:

* Patients who have undergone another form of bariatric surgery before RYGB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have scheduled a gastric bypass
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Medication use | one year
  Patients will be questioned preoperatively and one, three, six and twelve months after gastric bypass surgery. A questionnaire will be used to examine which drugs patients use and to what level they are adherent to treatment recommendations.

SECONDARY OUTCOMES:
Changes in dietary pattern before and after RYGB | one year
  The investigators will ask patients to keep a food record during two non-consecutive days preceding each consultation. In this food record patients have to note all consumed foods and beverages with the right/estimated amounts. This makes it possible to see changes of the composition of the meals before and after RYGB. The correlation between the dietary/total intake and clinical parameters will be investigated.
Medication counseling | one year
  Patients will be questioned preoperatively and one, three, six and twelve months after gastric bypass surgery. A questionnaire will be used to examine what kind of information they received about medication use pre- and post-RYGB.

CONTACTS AND LOCATIONS:
Overall Officials: Ina Gesquiere, PhD Student, Principal Investigator — Katholieke Universiteit Leuven - Centre for Pharmacotherapy; Veerle Foulon, Pharm PhD, Study Director — Katholieke Universiteit Leuven - Centre for Pharmacotherapy
Locations (1):
- KU Leuven - Centre for Pharmacotherapy, Leuven, Belgium